CLINICAL TRIAL: NCT01305863
Title: A Randomized, Controlled, Parallel Group, Blinded, Feasibility Study of the TGI Adipose-derived Stromal Cell (ASC)-Coated ePTFE Vascular Graft for Femoral-tibial Bypass Grafting.
Brief Title: Feasibility Study of the TGI Adipose-derived Stromal Cell (ASC)-Coated ePTFE Vascular Graft
Acronym: TGI-PVG-IDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tissue Genesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TGI-001-01-2008
Record Dates: First submitted 2011-02-10; First posted 2011-03-01 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Lower Limb Ischemia
Keywords: Peripheral Vascular Disease (PVD)
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propaten graft (Active Comparator): Untreated Propaten vascular graft
  Interventions: Device: Propaten graft
- ASC-Coated ePTFE graft (Experimental): ASC Coated BARD IMPRA® ePTFE Vascular Graft
  Interventions: Device: ASC coated ePTFE vascular graft

INTERVENTIONS:
Device: ASC coated ePTFE vascular graft — An ePTFE vascular graft in which the lumen of the graft has been coated with an autologous coating of adipose-derived stromal cells (ASC) prepared using an automated point-of-care processing instrument to facilitate isolation and concentration of autologous adipose-derived stromal cells and subsequent sodding of small-diameter vascular grafts.
  Other Names: TGI PVG
  Arms: ASC-Coated ePTFE graft
Device: Propaten graft — 6 mm Gore PROPATEN® graft (heparin-coated ePTFE vascular graft, thin-walled removable-ring stretch)
  Other Names: item HT060080A
  Arms: Propaten graft

SUMMARY:
Researchers are actively seeking a way to coat the inside of a synthetic graft so that it more closely resembles native vessels and therefore has low thrombogenicity and low incidence of stenosis. Using a biological coating comprised of autologous stromal cells derived from the patient's own adipose tissue is a logical solution. Considerable experimental evidence exists that such a coating is relatively non-thrombogenic and improves long-term graft patency.

The Company's TGI Cell Isolation System (CIS) for isolating and concentrating adipose-derived stromal cells (ASC) can be used to fill the pressing medical need for small-diameter synthetic vascular grafts. The TGI CIS enables the user to prepare a stem cell-based biological coating from adipose tissue liposuctioned from the patient. The cells derived from the adipose tissue are then sodded onto the internal lumen of the vascular graft to improve long term patency.

DETAILED DESCRIPTION:
Replacement or bypass of small diameter (< 4-5 mm) blood vessels is needed for a variety of medical problems, including peripheral vascular disease (PVD) associated with diabetes, generalized atherosclerosis, or aging), and critical limb ischemia (CLI). Vascular surgery has been extremely successful in replacing damaged or atherosclerotic arteries that are large in diameter and associated with high flow rates. However, as the diameter of the damaged vessel decreases, the ability to achieve long-term patency using replacement vessels decreases. The best current solution to this phenomenon of decreased patency with decreasing vessel diameter has been the use of the saphenous vein bypass graft. The saphenous vein has become the benchmark of all smaller diameter vascular grafts and demonstrates excellent patency when used from the femoral artery to the popliteal artery below the knee. However, when extended to more distal locations including the tibial arteries, even the saphenous vein begins to demonstrate limitations in its ability to maintain long-term patency.

The TGI ASC-coated expanded polytetrafluoroethylene (ePTFE) Vascular Graft is an adipose-derived stromal cell-sodded small-diameter vascular conduit intended for use as a peripheral bypass graft. The autologous cells used to create the ASC-coated vascular graft are isolated by the TGI Cell Isolation System (CIS). The TGI ASC-coated graft can be used to address the pressing medical need for small-diameter vascular grafts with improved long-term patency rates. The TGI CIS enables the user to prepare a stem cell-based biological coating in about an hour; stromal cells isolated from adipose tissue are sodded onto the internal lumen of the vascular graft before it is implanted into the patient during the course of a peripheral vascular bypass procedure.

The TGI Peripheral Vascular Graft (PVG) Kit consists of a vascular conduit, a proprietary enzymatic solution (Adipase™ Custom Enzyme Solution), and a disposable fluidics system, all to be used in conjunction with the TGI CIS, itself an automated point-of-care tissue processing instrument which isolates ASCs from a lipoaspirate specimen. Such cells are administered onto the lumen of the prepared conduit, a commercially available, small-diameter ePTFE straight vascular graft (IMPRA ePTFE Vascular Graft, item 80s06, Bard Peripheral Vascular, Inc.)

This instrument system will provide a sterile flow-path, through which cells are processed and separated. The flow-path is contained within a disposable cartridge that interlocks with the durable system hardware and includes both a flow-path cartridge with fluid reservoirs and a disposable centrifuge cartridge. The system is a self contained, stand-alone system requiring only AC power to operate.

The clinical trial process will involve a pilot (or feasibility) study to gain initial safety and effectiveness data in a limited human population. A subsequent pivotal study will be conducted with sufficient patient numbers to demonstrate a statistically significant improvement in effectiveness for defined clinical endpoints and to gain important safety information in a specific clinical population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old
2. Patient has a clinical diagnosis of Peripheral Vascular Disease (PVD) and requires a synthetic vascular graft, with the distal anastomosis to a tibial artery (peroneal, anterior tibial, posterior tibial).
3. The distal anastomosis must be no more distal than approximately the midcalf.
4. Rutherford-Baker classification for acute peripheral arterial disease of category 5 or less.
5. The proximal anastomosis must be in the common femoral artery (CFA) or the superficial femoral artery (SFA); the proximal anastomosis must not be above the inguinal ligament.
6. The distal target vessel must have continuous blood flow to the foot; an arteriovenous fistula must not be created at the distal anastomosis.

Exclusion Criteria:

1. Proximal anastomosis above the inguinal ligament.
2. Distal anastomosis below the mid-calf.
3. Lack of adequate subcutaneous fat stores to allow liposuction of 120 mL of adipose tissue.
4. Limb-threatening acute ischemia in the affected leg.
5. Active infection at the time of implantation.
6. Uncontrolled diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Graft patency | 6 months
  Graft patency will be measured by duplex ultrasound.

SECONDARY OUTCOMES:
Limb salvage | 12 months
  Amputation of limb or not
Wound Healing | 12 months
  Evidence of wound improvement
Rest Pain | 12 months
  Presence or absence of rest pain

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Morris, MD, Principal Investigator — The University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States